CLINICAL TRIAL: NCT02797470
Title: A Phase I Study of Stem Cell Gene Therapy for HIV Mediated by Lentivector Transduced, Pre-Selected CD34+ Cells
Brief Title: Gene Therapy in Treating Patients With Human Immunodeficiency Virus-Related Lymphoma Receiving Stem Cell Transplant
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-097; NCI-2015-01745 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9933 (Other: CTRP (Clinical Trial Reporting Program)); AMC 097 (Other: AIDS Malignancy Consortium); 097 (Other: AIDS Malignancy Consortium); AMC-097 (Other: CTEP); U01CA121947 (NIH)
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Results first posted 2023-07-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: HIV Infection; Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Plasmablastic Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Non-Hodgkin Lymphoma; Recurrent Burkitt Lymphoma; Recurrent Follicular Lymphoma; Stage III Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Follicular Lymphoma; Stage IV Mantle Cell Lymphoma
MeSH Terms: conditions — HIV Infections; Lymphoma, T-Cell; Plasmablastic Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — Carmustine; carmustine, poliferprosan 20 drug combination; Cytarabine; Etoposide; Melphalan; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (anti-HIV gene transduced CD34+ cells) (Experimental): Patients receive BEAM regimen administered as standard of care comprising carmustine on day -6, cytarabine BID on days -5 to -2, etoposide BID on days -5 to -2, and melphalan on day -1. Patients undergo infusion of lentivirus vector CCR5 shRNA/TRIM5alpha/TAR decoy-transduced autologous CD34-positive hematopoietic progenitor cells over 1 hour.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carmustine; Drug: Cytarabine; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Biological: Lentivirus Vector CCR5 shRNA/TRIM5alpha/TAR Decoy-transduced Autologous CD34-positive Hematopoietic Progenitor Cells; Drug: Melphalan; Procedure: Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo infusion of lentivirus vector CCR5 shRNA/TRIM5alpha/TAR decoy-transduced autologous CD34-positive hematopoietic progenitor cells
  Other Names: Autologous Stem Cell Transplantation
Drug: Carmustine — 300 mg/m2 on Day -6, as part of BEAM and R-BEAM regimens.
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; Gliadel; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Drug: Cytarabine — 100 mg/m2 BID on Days -5 through -2, as part of BEAM and R-BEAM regimens.
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Etoposide — VP-16: 100 mg/m2 BID on Days -5 through -2, as part of BEAM and R-BEAM regimens.
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Lentivirus Vector CCR5 shRNA/TRIM5alpha/TAR Decoy-transduced Autologous CD34-positive Hematopoietic Progenitor Cells — Undergo infusion of lentivirus vector CCR5 shRNA/TRIM5alpha/TAR decoy-transduced autologous CD34-positive hematopoietic progenitor cells
  Other Names: Lentivirus Vector CCR5 shRNA/TRIM5alpha/TAR Decoy-transduced Autologous CD34-positive HPCs
Drug: Melphalan — 140 mg/m2 on Day -1, as part of BEAM and R-BEAM regimens.
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo infusion of lentivirus vector CCR5 shRNA/TRIM5alpha/TAR decoy-transduced autologous CD34-positive hematopoietic progenitor cells
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation

SUMMARY:
This phase I/II trial studies the side effects and best dose of gene therapy in treating patients with human immunodeficiency virus (HIV)-related lymphoma that did not respond to therapy or came back after an original response receiving stem cell transplant. In gene therapy, small stretches of deoxyribonucleic acid (DNA) called "anti-HIV genes" are introduced into the stem cells in the laboratory to make the gene therapy product used in this study. The type of anti-HIV genes and therapy in this study may make the patient's immune cells more resistant to HIV-1 and prevent new immune cells from getting infected with HIV-1.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Safety, defined as timely engraftment (the collective establishment of a persistent absolute neutrophil count of at least 500 cells/mm^3 and platelet count of 20,000 cells/mm^3 without transfusion for 3 consecutive measurements of laboratory values obtained on different days) by one month post-transplant, in the absence of any grade 3 and 4 non-hematopoietic organ toxicity that can be attributed (possibly, probably, or definitely) to lentiviral transduced stem cell transplant, excluding alopecia, or any clonal expansion and excluding expected toxicities that are associated with the pre-transplant conditioning regimen.

SECONDARY OBJECTIVES:

I. To determine efficacy of the candidate product, defined as establishment of > 5% mononuclear blood cells expressing anti-HIV genes in the peripheral blood at 3 months post-transplant.

II. To determine the presence, quantity, and duration of gene modified HIV-1 resistant peripheral blood cells and gut mucosal immune cells.

III. To study the integration sites of vector sequences in circulating cells. IV. To study progression-free survival. V. To study overall survival. VI. To study complete response rate and duration. VII. To study partial response rate and duration. VIII. To study time to neutrophil engraftment (first measurement of 3 consecutive laboratory values on different days) of absolute neutrophil count [ANC] >= 500 cells/mm^3).

IX. To study time to platelet engraftment (first measurement of 3 consecutive measurements laboratory values obtained on different days) of platelets >= 20,000 cells/mm^3 without platelet transfusions 7 days prior).

X. To study hematologic function at day 100 (ANC > 1500, hemoglobin [Hb] > 10 g/dl without transfusion and platelets > 100,000) XI. To study CD4 recovery at the conclusion of the trial. XII. To study safety in terms of toxicities, infections, transfusions, and infusion-related reactions.

XIII. To study HIV-1 viral load over time. XIV. To study persistence of vector-transduced cells over time.

EXPLORATORY OBJECTIVE:

I. To evaluate the presence and the magnitude of expansion of HIV-1 resistant immune cells in the peripheral blood and gut mucosa of transplanted participants, subsequent to withholding anti-retroviral therapy (ART).

OUTLINE: This is a dose-escalation study of lentivirus vector CCR5 shRNA/TRIM5alpha/TAR decoy-transduced autologous CD34-positive hematopoietic progenitor cells.

Patients receive BEAM or BEAM-R regimen administered as standard of care comprising carmustine on day -6, cytarabine twice daily (BID) on days -5 to -2, etoposide BID on days -5 to -2, and melphalan on day -1. Patients with B-cell lymphoma also receive rituximab on day -6 before chemotherapy and on days 21 and 28 post-transplant as standard of care. Patients undergo intravenous (IV) infusion of lentivirus vector CCR5 shRNA/TRIM5alpha/TAR decoy-transduced autologous CD34-positive hematopoietic progenitor cells over 1 hour.

After completion of study treatment, patients are followed up at days 7, 14, 21, 28, 42, 60, 90, 120, 180, 240, 300, 360, 420, 480, 520, 600, 660, and 720, and then yearly for at least 15 years.

ELIGIBILITY:
Inclusion Criteria

* Inclusion criteria associated with type and status of lymphoma, one of the following must be applicable:

  * Biopsy-proven intermediate or high-grade non-Hodgkin's lymphoma, meeting one of the following criteria (timeline 8 months prior to enrollment in the screening segment):

    - In partial remission,

    - Relapsed after initial complete remission,

    - Failed induction therapy, but responds to salvage therapy (i.e., chemosensitive disease),

    - In complete remission with high-risk features as specified by the International Prognostic Index.
  * Biopsy-proven advanced stage follicular lymphoma, that have failed at least two lines of therapy multi-agent chemotherapy, but responds to salvage therapy i.e.,chemosensitive disease) (timeline 8 months prior to enrollment in the screening segment).
  * Biopsy-proven advanced stage Mantle cell lymphoma with Ki-67 > 10% in first complete remission (timeline 8 months prior to enrollment in the screening segment).
  * Biopsy-proven Hodgkin's lymphoma, meeting one of the following criteria (timeline 8 months prior to enrollment).

    - In first, or greater relapse after initial complete remission,

    - In partial remission,

    - Failed induction therapy, but responds to salvage therapy (i.e., chemosensitive disease).
  * Biopsy-proven Burkitt's lymphoma, meeting one of the following criteria (timeline 8 months prior to enrollment):

    - In second complete remission after relapse following initial complete remission,

    - Failed induction therapy, but responds (very good partial remission, complete remission, or near complete remission) to salvage therapy (i.e., chemosensitive disease).
  * Biopsy proven plasmablastic lymphomas, or peripheral T cell lymphoma (with the exception of ALK+ type in first or second complete remission) *NOTE: Patients meeting the following criteria are exempt from the 8-month timeline and do not require additional biopsy:

    * Patients who have never achieved a complete remission on the last biopsy-proven site of disease and went on to the next therapy then achieved a complete remission.
    * Patients who relapsed quickly (within 3 months of their last chemotherapy) and now have achieved a complete remission with salvage therapy.
* Inclusion criteria associated with HIV-1 status

  * HIV-1 infection, as documented by any federally approved, licensed HIV rapid test performed in conjunction with screening (or ELISA, test kit, and confirmed by Western blot or other approved test). Alternatively, this documentation may include a record demonstrating that another physician has documented the participant's HIV status based on either: 1) approved diagnostic tests, or 2) the referring physician's written record that HIV infection was documented, with supporting information on the participant's relevant medical history and/or current management of HIV infection.
  * Must be on a multi-drug anti-HIV regimen (excluding zidovudine [AZT, ZDV, Retrovir®, or agents containing zidovudine (e.g., Combivir® and Trizivir®)], and efavirenz [Sustiva®, or agents containing efavirenz (e.g., Atripla®)]).

Participants on zidovudine [AZT, ZDV, Retrovir®; including Combivir® and Trizivir®] and efavirenz [Sustiva®; including Atripla®] must switch to an alternative regimen without anticipated drug-drug interactions or myelosuppressive properties based on known viral resistance patterns and/or ART history, such as raltegravir and Truvada (emtricitabine and tenofovir) at least two weeks prior to the transplant.

o Participant taking ARTs must satisfy one of the following:

* Undetectable HIV viral load (< 50 copies/mL). For patients who have had negative viral loads in the past 6 months and no known HIV viral load >500 copies/mL within the last 6 months, minor fluctuations of viral load (isolated escalations up to 500 copies/mL) are acceptable. The participant's history of negative viral loads may be documented with recent laboratory results and/or a record from the participant's HIV care provider.
* If viral load is detectable at < 2000 copies/mL a review of previous antiretroviral regimens or previous genotypic or phenotypic testing which indicate the ability to fully suppress virus by addition of sensitive drugs must be performed. This review will be carried out by the protocol ID team or the ID specialist caring for the patient.
* If viral load is detectable at ≥ 2000 copies/mL, a current HIV genotype and/or phenotype must be obtained. If a HAART regimen to which the patient's virus is sensitive can be determined based on genotype and previous antiretroviral experience, then the patient will be considered eligible in this regard. This review will be carried out by the protocol ID team or the ID specialist caring for the patient.

General Inclusion Criteria (timeline: within 8 weeks prior to enrollment in the screening segment, unless otherwise specified)

* Karnofsky performance status of 70-100%. ECOG performance status <2
* SGOT and SGPT ≤ 2.5 times upper limit of normal (ULN). Serum bilirubin ≤ 2.5 times ULN except for participants who are on atazanavir or indinavir, or with elevated indirect bilirubin related to bilirubin conjugation issues such as Gilbert's disease, provided that the participant's direct bilirubin is within normal institutional limits.
* Participants who are hepatitis C virus antibody positive, or hepatitis B virus surface antigen positive must be free of clinical evidence of cirrhosis as determined by the principal investigator in consultation with the institutional Gastroenterology Service.
* Participants with Hepatitis B should be on appropriate anti-viral therapy at the time of the transplant, and their viral load should be negative.
* Serum creatinine ≤ 2 times ULN.
* Creatinine clearance ≥ 60 mL/min by the modified Cockcroft-Gault Formula.
* PT/PTT ≤ 2 times upper limit of normal (ULN), or international normalized ratio (INR)/PTT ≤ 2 times the ULN.
* FEV-1 or DLCO (corrected for hemoglobin) ≥ 50% predicted.
* LVEF ≥ 50% by 2D ECHO or MUGA scan.
* Not pregnant or nursing, with negative serum pregnancy test. Pregnant women are excluded from this study because the conditioning regimen has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with BEAM, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study.
* Participants should agree to practice effective contraceptive precautions and to use at least one method of contraception for the duration of the study and for 3 months post-transplant.
* Age ≥18 years. Because only adult transplant centers are participating as study sites.

  * Life expectancy of greater than 3 months.
  * Ability to understand and the willingness to sign a written informed consent document.
  * Receipt of a stable ART regimen for at least 3 weeks prior to enrollment.

Exclusion Criteria

Participants who do not fulfill the criteria as listed above, are ineligible. Additionally, the presence of any of the following conditions will exclude a participant from study enrollment (timeline for all the exclusion criteria is within 8 weeks prior to enrollment in the screening segment):

* Participants with > 5% involvement of bone marrow by malignant cells (either by manual count or flow cytometry) prior to stem cell collection.
* Participants with any abnormal cytogenetics in the bone marrow not related to the lymphoma, and not deemed to be constitutional.
* Participants with unexplained anemia and/or thrombocytopenia.
* Participants with clear evidence of myeloproliferative disorders, or myelodysplastic disorders in the marrow.
* Presence of any active CNS disease at the time of evaluation (parenchymal or leptomeningeal).
* Any history of HIV-1 associated encephalopathy.
* Participants with persistently low CD4 counts less than 200 and a history of any AIDS-defining infection in the last 6 months before screening are excluded from the study.
* Symptomatic/active bacterial, or fungal, or any other opportunistic infection.
* Active CMV retinitis, or other active CMV-related organ dysfunction.
* Relapse of pneumocystis carinii pneumonia within the past year before enrollment.
* Intractable, severe diarrhea, defined as > 1.500 cc diarrheal fluid per day, or diarrhea causing persistent severe electrolyte abnormalities, or hypoalbuminemia.
* History of active myocardial ischemia, cardiomyopathy, uncontrolled dysrhythmia, or congestive heart failure within the last 6 months before enrollment.
* Dementia of any kind.
* Seizures within the past 12 months before enrollment.
* History of Grade III hemorrhagic cystitis due to prior cyclophosphamide chemotherapy.
* History of other prior malignancy, except squamous cell carcinoma of the cervix or anus, superficial basal cell or squamous cell skin cancer, or other malignancy curatively treated more than 5 years ago before enrollment.
* Active psychosocial condition that would hinder study compliance and follow-up.
* Any perceived inability to directly (and without the means of a legal guardian) provide informed consent.
* Any medical or physical contraindication, or other inability to undergo HPC collection.
* Participants who are receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2036-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Abedi, Principal Investigator — AIDS Malignancy Consortium
Locations (4):
- United States (4):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: Patients receive BEAM regimen administered as standard of care comprising carmustine on day -6, cytarabine BID on days -5 to -2, etoposide BID on days -5 to -2, and melphalan on day -1. Patients undergo infusion of lentivirus vector CCR5 shRNA/TRIM5alpha/TAR decoy-transduced autologous CD34-positive hematopoietic progenitor cells over 1 hour.
  Autologous Hematopoietic Stem Cell Transplantation: Undergo infusion of lentivirus vector CCR5 shRNA/TRIM5alpha/TAR decoy-transduced autologous CD34-positive hematopoietic progenitor cells
  Carmustine: 300 mg/m2 on Day -6, as part of BEAM and R-BEAM regimens.
  Cytarabine: 100 mg/m2 BID on Days -5 through -2, as part of BEAM and R-BEAM regimens.
  Etoposide: VP-16: 100 mg/m2 BID on Days -5 through -2, as part of BEAM and R-BEAM regimens.
  Laboratory Biomarker Analysis: Correlative studies
  Lentivirus Vector CCR5 shRNA/TRIM5alpha/TAR Decoy-transduced Autologous CD34-positive Hematopoietic Progenitor Cells: Undergo infusion of lentivirus vector CCR5 shRNA/TRIM5alpha/TAR decoy-transduced autologous CD34-positive hematopoietic progenitor cells
  Melphalan: 140 mg/m2 on Day -1, as part of BEAM and R-BEAM regimens.
  Peripheral Blood Stem Cell Transplantation: Undergo infusion of lentivirus vector CCR5 shRNA/TRIM5alpha/TAR decoy-transduced autologous CD34-positive hematopoietic progenitor cells
- Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio; Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: Patients receive BEAM regimen administered as standard of care comprising carmustine on day -6, cytarabine BID on days -5 to -2, etoposide BID on days -5 to -2, and melphalan on day -1. Patients undergo infusion of lentivirus vector CCR5 shRNA/TRIM5alpha/TAR decoy-transduced autologous CD34-positive hematopoietic progenitor cells over 1 hour.
  Autologous Hematopoietic Stem Cell Transplantation: Undergo infusion of lentivirus vector CCR5 shRNA/TRIM5alpha/TAR decoy-transduced autologous CD34-positive hematopoietic progenitor cells
Period: Overall Study
Arm/Group | Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio | Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio | Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio
Started | 5 | 4 | 2
Completed | 5 | 4 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants received Stem Cell Gene Therapy
Arm/Group | Treatment (Anti-HIV Gene Transduced CD34+ Cells)
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Patients per arm were displayed.
  years
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: number analyzed (Participants) | 5
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio | 61 (6.4)
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: number analyzed (Participants) | 4
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio | 51 (4.7)
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: number analyzed (Participants) | 2
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio | 61 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Patients per arm were displayed.
  Participants
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: number analyzed (Participants) | 5
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: Female | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: Male | 5
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: number analyzed (Participants) | 4
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: Female | 1
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: Male | 3
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: number analyzed (Participants) | 2
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: Female | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Patients per arm were displayed.
  Participants
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: number analyzed (Participants) | 5
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: Hispanic or Latino | 1
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: Not Hispanic or Latino | 4
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: Unknown or Not Reported | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: number analyzed (Participants) | 4
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: Hispanic or Latino | 1
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: Not Hispanic or Latino | 3
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: Unknown or Not Reported | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: number analyzed (Participants) | 2
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: Hispanic or Latino | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: Not Hispanic or Latino | 2
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Patients per arm were displayed.
  Participants
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: number analyzed (Participants) | 5
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: American Indian or Alaska Native | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: Asian | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: Native Hawaiian or Other Pacific Islander | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: Black or African American | 1
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: White | 3
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: More than one race | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: Unknown or Not Reported | 1
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: number analyzed (Participants) | 4
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: American Indian or Alaska Native | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: Asian | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: Native Hawaiian or Other Pacific Islander | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: Black or African American | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: White | 3
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: More than one race | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: Unknown or Not Reported | 1
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: number analyzed (Participants) | 2
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: American Indian or Alaska Native | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: Asian | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: Native Hawaiian or Other Pacific Islander | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: Black or African American | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: White | 2
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: More than one race | 0
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: Unknown or Not Reported | 0
Bone Marrow Biopsy status [Count of Participants; unit: Participants] — Population: Patients per arm were displayed.
  Participants
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio: number analyzed (Participants) | 5
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio | 4
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio: number analyzed (Participants) | 4
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio | 4
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio: number analyzed (Participants) | 2
    Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve a Timely Engraftment
Description: Timely engraftment is defined as a persistent an absolute neutrophil count (ANC) of at least 500 cells/mm3 and a platelet count of at least 20,000 cells/mm3 for at least 3 days
Time Frame: 1 month post-transplant
Measure: Mean (95% Confidence Interval); unit: percentage of participants who achieve a
Arm/Group | Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio | Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio | Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio
Number analyzed (Participants) | 5 | 4 | 2
percentage of participants who achieve a | 60 [14.7 to 94.7] | 75 [19.4 to 99.4] | 100 [15.8 to 100]

2. Secondary Outcome: Proportion of Study Participants Who Achieve Greater Than 5% Mononuclear Blood Cells Expressing Anti-HIV Genes in Peripheral Blood
Description: To determine efficacy of the candidate product, defined as establishment of > 5% mononuclear blood cells expressing anti-HIV genes
Time Frame: 3 months post-transplant
Reporting Status: Not Posted

3. Secondary Outcome: Proportion of Study Participants With Gene Modified HIV-1 Resistant Peripheral Blood Cells and Gut Mucosal Immune Cells
Description: To determine the presence, quantity, and duration of gene modified HIV-1 resistant peripheral blood cells and gut mucosal immune cells
Time Frame: Up to 24 months post-transplant
Reporting Status: Not Posted

4. Secondary Outcome: Quantity of Gene Modified HIV-1 Resistant Peripheral Blood Cells and Gut Mucosal Immune Cells
Description: Summarized descriptively. Continuous measures will be summarized by mean (standard deviation [SD]) and median (range), with log transformation if necessary for skewed measures, as would be typical for cell counts.
Time Frame: Up to 24 months post-transplant
Reporting Status: Not Posted

5. Secondary Outcome: Integration Sites of Vector Sequences in Circulating Cells
Description: Single genome sequencing of HIV gp120 and HIV pol will be performed to understand sequence evolution following transplantation and detection of minority resistance variants.
Time Frame: Up to 24 months post-transplant
Reporting Status: Not Posted

6. Secondary Outcome: Progression-free Survival
Description: Time-to-event data will be presented graphically by Kaplan-Meier plots and summarized by estimated median time to event (if that is estimable from the data) with 95% confidence interval.
Time Frame: Time from start of study treatment to relapse, progression, or death from any cause
Reporting Status: Not Posted

7. Secondary Outcome: Overall Survival
Description: The length of time from the start of treatment until death
Time Frame: Up to 15 years
Reporting Status: Not Posted

8. Secondary Outcome: Number of Participants With a Complete Response
Description: A complete response is the complete disappearance of any disease, as determined by imaging
Time Frame: 24 months
Reporting Status: Not Posted

9. Secondary Outcome: Number of Days From the First Documentation of a Complete Response Until the First Day of Relapse
Description: Complete response is defined as the absence of any disease on imaging or by exam; progressive disease is defined as new lesions or new evidence of disease
Time Frame: Time from the first documentation of CR until first date that relapsed or progressive disease is objectively documented, assessed up to 15 years
Reporting Status: Not Posted

10. Secondary Outcome: Partial Response Rate and Duration
Description: Will be assessed following the Lugano Classification. In the absence of evident disease progression, response will be assessed formally at 3, 6, 12 and 24 months post transplant per study calendar.
Time Frame: Up to 15 years
Reporting Status: Not Posted

11. Secondary Outcome: Time to Neutrophil Engraftment
Description: First measurement of 3 consecutive laboratory values obtained on different days) of ANC > 500 cells/mm3
  .
Time Frame: Up to 15 years
Reporting Status: Not Posted

12. Secondary Outcome: Time to Platelet Engraftment
Description: First measurement of 3 consecutive laboratory values obtained on different days) of platelets > 20,000 cells/mm3 without platelet transfusions 7 days prior
Time Frame: Up to 15 years
Reporting Status: Not Posted

13. Secondary Outcome: Number of Participants With an Absolute Neutrophil Count of at Least 1500 Cells/mm3, Hemoglobin of at Least 10 g/dL, and Platelets Greater Than 100,000.
Description: To study hematologic function at Day 100
Time Frame: 100 days
Reporting Status: Not Posted

14. Secondary Outcome: CD4 Count Recovery
Description: At six months post-transplant, or later, ART will be voluntarily withheld for a 12 week period only for participants who have a CD4 count of 300 or higher with no detectable viral load. for participants in which the CD4 T-cell count has not risen to ≥ 300 cells/mm3 at the time of the planned ART interruption, ART will continue until the T-cell count has risen to ≥ 300 cells/mm3.
Time Frame: Up to 24 months post-treatment
Reporting Status: Not Posted

15. Secondary Outcome: Number of Participants With Adverse Events as Assessed by the CTCAE
Description: To study safety in terms of the frequency of toxicities, infections, transfusions, and infusion-related reactions
Time Frame: Up to 15 years
Reporting Status: Not Posted

16. Secondary Outcome: HIV-1 Viral Load
Description: To study HIV-1 viral load over time
Time Frame: At week 4, months 3, 6, 8, 10, 12, 14, 16, 20, and 24 post-transplant.
Reporting Status: Not Posted

17. Secondary Outcome: Persistence of Vector-transduced Cells Over Time
Description: Vector stability analysis will be performed via qPRC sequencing.
Time Frame: Up to 15 years
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Expansion of HIV-1 Resistant Immune Cells
Description: Presence and the magnitude of expansion of HIV-1 resistant immune cells in the peripheral blood and gut mucosa of transplanted participants, subsequent to withholding ART
Time Frame: Up to 24 months post-transplant
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 months after transplant
Arm/Group | Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio | Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio | Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio
All-Cause Mortality (participants affected / at risk) | 2/5 | 2/4 | 1/2
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/4 | 0/2
Other Adverse Events (participants affected / at risk) | 2/5 | 4/4 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio (N=5) | Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio (N=4) | Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio (N=2)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:0 Ratio (N=5) | Treatment (Anti-HIV Gene Transduced CD34+ Cells): 1:1 Ratio (N=4) | Treatment (Anti-HIV Gene Transduced CD34+ Cells): 5:1 Ratio (N=2)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 (2) | 2 (2) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 2 (2) | 0 (0)
WHITE BLOOD CELL DECREASED (Investigations) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT02797470/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT02797470/ICF_001.pdf